CLINICAL TRIAL: NCT02333487
Title: Interventional, Open-label, Positron Emission Tomography (PET) Study Investigating D1 Dopamine, D2 Dopamine, and 5-HT6 Serotonin Receptor Occupancy After Multiple Oral Dosing of Lu AF35700 in Male Patients With Schizophrenia
Brief Title: Positron Emission Tomography (PET) Study Investigating Dopamine and Serotonin Receptor Occupancy After Multiple Oral Dosing of Lu AF35700
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15859A
Record Dates: First submitted 2015-01-06; First posted 2015-01-07 (Estimated); Results first posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Lu AF35700

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lu AF35700 (Group D1) (Experimental): Up to 3 PET scans, besides baseline scan, using [11C]-NNC 112 tracer to detect D1 dopamine receptor occupancy before and after multiple oral dosing of Lu AF35700
  Interventions: Drug: Lu AF35700
- Lu AF35700 (Group D2) (Experimental): Up to 3 PET scans, besides baseline scan, using [11C]-Raclopride to detect D2 dopamine receptor occupancy before and after multiple oral dosing of Lu AF35700
  Interventions: Drug: Lu AF35700
- Lu AF35700 (Group 5-HT6) (Experimental): Up to 3 PET scans, besides baseline scan, using [11C]- Lu AE60157 tracer to detect 5-HT6 (5-hydroxytryptamine-6) receptor occupancy before and after multiple oral dosing of Lu AF35700
  Interventions: Drug: Lu AF35700

INTERVENTIONS:
Drug: Lu AF35700 — 5 mg tablets for oral administration

SUMMARY:
The purpose of this PET study is to verify the binding of Lu AF35700 after multiple oral dosing at the dopamine and the serotonin receptors in male patients with schizophrenia.

DETAILED DESCRIPTION:
There were 3 to 4 cohorts of 2 patients per receptor group. Lu AF35700 was administered as multiple oral doses for up to 21 days before the PET scans were performed. The doses in all groups were selected with the aim of characterising the exposure response (occupancy) curve. The doses for all groups, with the exception of A1, B1, and C1, were subject to change within the dose range already investigated and found tolerable. The next dose for the groups was established at a dosing conference based on an evaluation of the occupancy obtained, and safety, tolerability, and pharmacokinetic data from all previous cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is a man aged between ≤18 and ≥60 years
2. BMI of ≥19 kg/m2 to ≤ 37 kg/m2
3. The patient has a primary diagnosis of schizophrenia according to DSM-5™ (code 295.90)
4. The patient has a Clinical Global Impression - Severity of Illness (CGI-S) score ≤ 4 (moderately ill) at screening and safety baseline
5. The patient is currently under oral therapy with one or more of the antipsychotic medications listed in Appendix II.
6. The patient has a Positive and Negative Syndrome Scale (PANSS) total score ≤ 80
7. The patient has a score of ≤ 4 (moderate) on the following PANSS items at screening and at safety baseline: P7 (hostility), G8 (uncooperativeness)

Exclusion Criteria:

1. The patient experienced an acute exacerbation requiring hospitalization within the last 3 months.
2. The patient experienced an acute exacerbation requiring change in antipsychotic medication (with reference to drug or dose) within the last 4 weeks.
3. The patient has a diagnosis or history of substance use disorder (except nicotine) according to DSM-5-TR® criteria ≤3 months prior to screening
4. The patient is at significant risk of harming himself or others according to the investigator's judgment or as indicated by an answer of "yes" to the question 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) at the Screening Visit within the last six months on the lifetime version of C-SSRS.
5. Based on investigators judgment the patient has a medical or neurological disorder or treatment for such disorder that could interfere with the study treatment or impair treatment compliance.
6. The patient has had past episodes of extrapyramidal symptoms (EPS) under current medication within the last 3 month
7. The patient takes other medication than those listed as allowed concomitant medication in Appendix III
8. The patient is occupationally exposed to significant levels of ionizing radiation.

Other protocol-defined inclusion and exclusion criteria may apply

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2014-12-30 (Actual); Primary Completion 2016-02-11 (Actual); Study Completion 2016-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (1):
- US802, Rockville, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of 6 to 8 patients assigned to one of 3 groups (D1, D2, or 5-HT6). Each group characterising the Lu AF35700 plasma concentration/receptor occupance (RO) relationship of 1 of 3 receptors using 1 of 3 ligands: Group D1 using [11C]-NNC 112, Group D2 using [11C]-raclopride, and Group 5-HT6 using [11C]-Lu AE60157
Groups:
- Lu AF35700 (Group D1): Lu AF35700: Daily dosing for up to 21 days (10 mg for 21 days for Cohort A1, 10 mg for 3 days and 15 mg for 18 days for Cohort A2, and 10 mg for 3 days and 20 mg for 17 days for Cohort A3).
  D1 receptor occupancy measured using [11C]-NNC 112.
- Lu AF35700 (Group D2): Lu AF35700: Daily dosing for 21 days (10 mg for 3 days and 20 mg for 18 days).
  D2 receptor occupancy measured using [11C]-raclopride.
- Lu AF35700 (Group 5-HT6): Lu AF35700: Cohort C1: Daily dosing with 10 mg for 21 days, Cohort C2: Daily dosing with 5 mg for 21 days, Cohort C3: Daily dosing with 5 mg for 7 days, Cohort C4: Dosing with 5 mg for 4 days (Days 1, 3, 5, and 7).
  5-HT6 receptor occupancy measured using [11C]-Lu AE60157.
Period: Overall Study
Arm/Group | Lu AF35700 (Group D1) | Lu AF35700 (Group D2) | Lu AF35700 (Group 5-HT6)
Started | 6 | 8 | 8
Completed | 6 | 6 | 8
Not Completed | 0 | 2 | 0
Not completed — Adverse Event | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Lu AF35700 (Group 5-HT6): Lu AF35700: Cohort C1: Daily dosing with 10 mg for 21 days, Cohort C2: Daily dosing with 5 mg for 21 days, Cohort C3: Daily dosing with 5 mg for 7 days, and Cohort C4: Dosing with 5 mg for 4 days (Days 1, 3, 5, and 7).
  5-HT6 receptor occupancy measured using [11C]-Lu AE60157.
- Total: Total of all reporting groups
Arm/Group | Lu AF35700 (Group D1) | Lu AF35700 (Group D2) | Lu AF35700 (Group 5-HT6) | Total
Number analyzed (Participants) | 6 | 8 | 8 | 22
Age, Continuous [Mean (Full Range); unit: years] | 41 [28 to 59] | 39 [27 to 52] | 43 [28 to 57] | 41 [27 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 6 | 8 | 8 | 22
Region of Enrollment [Number; unit: participants]
  United States | 6 | 8 | 8 | 22

OUTCOME MEASURES:

1. Primary Outcome: Emax D1 Dopamine
Description: Maximal target occupancy (Emax) on the D1 dopamine receptor using PET with [11C]-NNC 112 tracer compound.
  The relationship between systemic exposure of Lu AF35700 and D1 dopamine occupancy was investigated using an Emax model containing the regression parameters maximal target occupancy (Emax) and plasma concentration which gives 50% of Emax (EC50). Both Emax and EC50 were estimated using one model for all post-baseline scans combined. No statistical testing was performed.
Time Frame: Change from baseline to 344 hours post last dose
Measure: Number (95% Confidence Interval); unit: percentage
Groups:
- Lu AF35700 (Group D1): Lu AF35700: Daily dosing for up to 21 days (10 mg for 21 days for Cohort A1, 10 mg for 3 days and 15 mg for 18 days for Cohort A2, and 10 mg for 3 days and 20 mg for 17 days for Cohort A3).
Arm/Group | Lu AF35700 (Group D1)
Number analyzed (Participants) | 6
percentage | 81.9 [73.5 to 90.4]

2. Primary Outcome: EC50 D1 Dopamine
Description: Plasma concentration which gives 50% of Emax (EC50)
  The relationship between systemic exposure of Lu AF35700 and D1 dopamine occupancy was investigated using an Emax model containing the regression parameters maximal target occupancy (Emax) and plasma concentration which gives 50% of Emax (EC50). Both Emax and EC50 were estimated using one model for all post-baseline scans combined. No statistical testing was performed.
Time Frame: Change from baseline to 344 hours post last dose
Measure: Number (95% Confidence Interval); unit: ng/mL
Arm/Group | Lu AF35700 (Group D1)
Number analyzed (Participants) | 6
ng/mL | 1.4 [0.8 to 2.0]

3. Primary Outcome: Emax D2 Dopamine
Description: Maximal target occupancy (Emax) on the D2 dopamine receptor using PET with [11C]-Raclopride tracer compound.
  The relationship between systemic exposure of Lu AF35700 and D2 dopamine occupancy was investigated using an Emax model containing the regression parameters maximal target occupancy (Emax) and plasma concentration which gives 50% of Emax (EC50). Emax was estimated using one model for all post-baseline scans combined. No statistical testing was performed.
Time Frame: Change from baseline to 344 hours post last dose
Measure: Number; unit: percentage
Groups:
- Lu AF35700 (Group D2): Lu AF35700: Daily dosing for 21 days (10 mg for 3 days and 20 mg for 18 days)
Arm/Group | Lu AF35700 (Group D2)
Number analyzed (Participants) | 8
percentage | 102

4. Primary Outcome: EC50 D2 Dopamine
Description: Plasma concentration which gives 50% of Emax (EC50)
  The relationship between systemic exposure of Lu AF35700+Lu AF36152 and D2 dopamine occupancy was investigated using an Emax model containing the regression parameters maximal target occupancy (Emax) and plasma concentration which gives 50% of Emax (EC50). Both Emax and EC50 were estimated using one model for all post-baseline scans combined. No statistical testing was performed.
Time Frame: Change from baseline to 344 hours post last dose
Measure: Number (95% Confidence Interval); unit: ng/mL
Arm/Group | Lu AF35700 (Group D2)
Number analyzed (Participants) | 8
ng/mL | 29.1 [15.9 to 42.4]

5. Primary Outcome: Emax 5-HT6 Serotonin
Description: Maximal target occupancy (Emax) on the 5-HT6 receptor using PET with [11C]-Lu AE60157 as tracer compound.
  The relationship between systemic exposure of Lu AF35700+Lu AF36152 and 5-HT6 occupancy was investigated using an Emax model containing the regression parameters maximal target occupancy (Emax) and plasma concentration which gives 50% of Emax (EC50). Emax was estimated using one model for all post-baseline scans combined. No statistical testing was performed.
Time Frame: Change from baseline to 344 hours post last dose
Measure: Number (95% Confidence Interval); unit: percentage
Groups:
- Lu AF35700 (Group 5-HT6): Lu AF35700: Cohort C1: Daily dosing with 10 mg for 21 days, Cohort C2: Daily dosing with 5 mg for 21 days, Cohort C3: Daily dosing with 5 mg for 7 days, and Cohort C4: Dosing with 5 mg for 4 days (Days 1, 3, 5, and 7).
Arm/Group | Lu AF35700 (Group 5-HT6)
Number analyzed (Participants) | 8
percentage | 88.1 [84.1 to 92.1]

6. Primary Outcome: EC50 5-HT6 Serotonin
Description: Plasma concentration which gives 50% of Emax (EC50)
  The relationship between systemic exposure of Lu AF35700+Lu AF36152 and 5_HT6 serotonin occupancy was investigated using an Emax model containing the regression parameters maximal target occupancy (Emax) and plasma concentration which gives 50% of Emax (EC50). Both Emax and EC50 were estimated using one model for all post-baseline scans combined. No statistical testing was performed.
Time Frame: Change from baseline to 344 hours post last dose
Measure: Number (95% Confidence Interval); unit: ng/mL
Arm/Group | Lu AF35700 (Group 5-HT6)
Number analyzed (Participants) | 8
ng/mL | 0.4 [0.2 to 0.5]

ADVERSE EVENTS:
Time Frame: Up to week 12.
Description: Adverse Events were monitored irrespective of Lu AF35700 dosing cohort, i.e., unable to know what Lu AF35700 dose event occurred at.
  It was pre-specified in the study to report Adverse Events by tracer group only.
Groups:
- Lu AF35700 (Group D1): Lu AF35700: Daily dosing for up to 21 days (10 mg for 21 days for Cohort A1, 10 mg for 3 days and 15 mg for 18 days for Cohort A2, and 10 mg for 3 days and 20 mg for 17 days for Cohort A3).
  D1 receptor occupancy using [11C]-NNC 112
- Lu AF35700 (Group D2): Lu AF35700: Daily dosing for 21 days (10 mg for 3 days and 20 mg for 18 days).
  D2 receptor occupancy using [11C]-raclopride
- Lu AF35700 (Group 5-HT6): Lu AF35700: Cohort C1: Daily dosing with 10 mg for 21 days, Cohort C2: Daily dosing with 5 mg for 21 days, Cohort C3: Daily dosing with 5 mg for 7 days, and Cohort C4: Dosing with 5 mg for 4 days (Days 1, 3, 5, and 7).
  5-HT6 (5-hydroxytryptamine-6) receptor occupancy using [11C]-Lu AE60157
Arm/Group | Lu AF35700 (Group D1) | Lu AF35700 (Group D2) | Lu AF35700 (Group 5-HT6)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/6 | 1/8 | 1/8
Other Adverse Events (participants affected / at risk) | 5/6 | 6/8 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lu AF35700 (Group D1) (N=6) | Lu AF35700 (Group D2) (N=8) | Lu AF35700 (Group 5-HT6) (N=8)
Chest pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Worsening of schizophrenia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lu AF35700 (Group D1) (N=6) | Lu AF35700 (Group D2) (N=8) | Lu AF35700 (Group 5-HT6) (N=8)
Anxiety (Psychiatric disorders) | 2 (4) | 2 (6) | 1 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Psychotic Disorder (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 2 (12) | 3 (7) | 2 (2)
Tympanic Membrane Disorder (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Blood Urine Present (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight Increased (Investigations) | 1 (1) | 3 (3) | 2 (2)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Schizophrenia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Tootache (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotarnsferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyl transferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Axillary mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Penis disorder (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
An estimate of the confidence interval for the parameter Emax in the dopamine D2 receptor occupancy model was not calculable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No